CLINICAL TRIAL: NCT04724928
Title: Evaluating the Impact of 18F-FDG-PET-CT on Risk Stratification and Treatment Adaptation for Patients with Muscle Invasive Bladder Cancer (EFFORT-MIBC): a Phase II Prospective Trial
Brief Title: Evaluating the Impact of 18F-FDG-PET-CT on Risk Stratification and Treatment Adaptation for Patients with Muscle Invasive Bladder Cancer
Acronym: EFFORT-MIBC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Kom Op Tegen Kanker (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC-07456; BC-07456 (Other: Ethics committee of the Ghent University Hospital)
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Muscle-Invasive Bladder Carcinoma
Keywords: 18F-FDG-PET-CT; Staging; Distand metastasis; Oligometastatic disease; Metastasis directed therapy; Immunotherapy
MeSH Terms: interventions — Immunotherapy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Non-metastatic MIBC (Active Comparator): No signs of extra-pelvic metastasis on conventional imaging (abdominopelvic and thoracic CT/MRI) and 18F-FDG-PET-CT's
  Interventions: Procedure: Standard of care
- Oligo-metastatic MIBC on 18F-FDG-PET-CT (Experimental): No signs of extra-pelvic metastasis on conventional imaging (abdominopelvic and thoracic CT/MRI) but presence of ≤ 3 metastasis on 1 or both 18F FDG PET-CT 's
  Interventions: Radiation: Metastasis directed therapy (MDT)
- Poly-metastatic MIBC on 18F-FDG-PET-CT (Experimental): No signs of extra-pelvic metastasis on conventional imaging (abdominopelvic and thoracic CT/MRI) but presence of > 3 metastasis on 1 or both 18F FDG PET-CT 's
  Interventions: Drug: Immunotherapy

INTERVENTIONS:
Radiation: Metastasis directed therapy (MDT) — Patient receives standard of care therapy with either radical cystectomy with pelvic lymph node dissection or trimodality therapy (consisting of a visible complete TURb and radio chemotherapy). Concurrently, the oligometastasis will be treated with stereotactic body radiotherapy or metastasectomy.
  Arms: Oligo-metastatic MIBC on 18F-FDG-PET-CT
Drug: Immunotherapy — Patient receives standard of care therapy with either radical cystectomy with pelvic lymph node dissection or trimodality therapy (consisting of a visible complete TURb and radio chemotherapy). Afterwards immunotherapy will be initiated and regular follow up will be performed.
  Arms: Poly-metastatic MIBC on 18F-FDG-PET-CT
Procedure: Standard of care — Patient receives standard of care therapy with either radical cystectomy with pelvic lymph node dissection or trimodality therapy (consisting of a visible complete TURb and radio chemotherapy). Afterwards regular follow up is performed.
  Arms: Non-metastatic MIBC

SUMMARY:
Evaluate the impact of 18F-FDG-PET-CT on the staging of patients with muscle invasive bladder cancer. Based on the results of 2 18F-FDG-PET-CT's patients are stratified in non-metastatic, oligometastatic and polymetastatic bladder cancer patients and the treatment is adapted accordingly to improve overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Histopathology-proven MIBC on TURb or ≥ T3 on conventional imaging treated with MIBC radical treatment
* T1-4 N0-3 M0 MIBC on conventional imaging (thoracic CT and abdominopelvic CT/ MRI)
* Age > 18 years
* WHO 0-2
* Willingness to undergo 18F-FDG-PET-CT
* Willingness to undergo MDT or immunotherapy, in case of diagnosis of oligometastatic or polymetastatic disease on 18F-FDG-PET-CT, respectively
* Willingness and ability to provide a signed informed consent according to ICH/GCP and national/local regulations

Exclusion Criteria:

* Presence of distant metastasis on conventional imaging (thoracic CT and abdominopelvic CT/ MRI)
* Refusal of or having contraindications to 18F-FDG-PET-CT
* Refusal of MDT or immunotherapy
* Prior radiotherapy unabling MDT
* Contraindications to radiotherapy (including active inflammatory bowel disease)
* Contraindications to immunotherapy
* Other primary tumor diagnosed < 5 years ago and for which treatment is still required, except for diagnosis of non-metastatic prostate cancer at time of diagnosis of MIBC or non-melanoma skin cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
  Defined as the time from diagnosis of MIBC to death from any cause

SECONDARY OUTCOMES:
The number of patients with acute toxicity | 3 months
  Assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0
The number of patients with late toxicity | 5 years
  Assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Progression-free survival | 5 years
  Defined as appearance of local/locoregional recurrence diagnosed at CT-scan or cystoscopy in case of TMT or appearance of metastasis diagnosed at MIBC or non-MIBC-related imaging.
Distant metastasis-free survival | 5 years
  Defined as time of diagnosis until occurrence of distant metastasis on repeated imaging.
Disease specific survival | 5 years
  Defined as time of diagnosis until death due to MIBC.
Patient reported quality of life as per EORTC-QLQ C30 | 5 years
  Validated questionnaire assessing different health-related parameters (psychological, physical and social well-being) in cancer patients
Patient reported quality of life as per EORTC-QLQ BLM30 | 5 years
  Validated questionnaire assessing the health-related QOL of muscle invasive bladder cancer patients
Sensitivity/specificity of 18F-FDG-PET-CT for the detection of extra-pelvic metastases | 3 months
  Sensitivity/specificity of 18F-FDG-PET-CT
Validation of predictive biomarkers | 5 years
  A biopsy specimen of the bladder, obtained after transurethral resection of the bladder (TURb),as well as urine and blood samples will be collected for validation of predictive biomarkers by evaluating the correlation between response to therapy and outcome (PFS, DMFS, DSS and OS) with in literature reported biomarkers determined on biopsy specimen of the bladder, obtained after TURb.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Fonteyne, MD; PhD, Principal Investigator — UZ Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verghote F, Poppe L, Verbeke S, Dirix P, Albersen M, De Meerleer G, Berghen C, Ost P, Villeirs G, De Visschere P, De Man K, De Maeseneer D, Rottey S, Van Praet C, Decaestecker K, Fonteyne V. Evaluating the impact of 18F-FDG-PET-CT on risk stratification and treatment adaptation for patients with muscle-invasive bladder cancer (EFFORT-MIBC): a phase II prospective trial. BMC Cancer. 2021 Oct 18;21(1):1113. doi: 10.1186/s12885-021-08861-x. PMID 34663254